CLINICAL TRIAL: NCT00699712
Title: Multi-Center, Open Label, Dose Escalating, Sequential Group Study to Assess the Hemodynamic Effects, Safety and Tolerability of CD-NP in Patients With Stabilized Acute Heart Failure (AHF)
Brief Title: Study to Assess Hemodynamic Effects, Safety and Tolerability of Chimeric Natriuretic Peptide (CD-NP) in Patients With Stabilized Acute Heart Failure (AHF)
Acronym: PreCONDITION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nile Therapeutics (Industry)
Collaborators: Momentum Research, Inc. (Industry)
Responsible Party: Hsiao Lieu, MD / Vice President, Clinical Research, Nile Therapeutics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIL-CDNP-CT003
Record Dates: First submitted 2008-06-10; First posted 2008-06-18 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ADHF; AHF; HF
MeSH Terms: interventions — cenderitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Open-label regimen of doses 1 and 2 of CDNP
  Interventions: Drug: CD-NP (Chimeric natriuretic peptide)
- B (Experimental): Open-label regimen of doses 2 and 3 of CDNP
  Interventions: Drug: CD-NP (Chimeric natriuretic peptide)
- C (Experimental): Open-label regimen of doses 3 and 4 of CDNP
  Interventions: Drug: CD-NP (Chimeric natriuretic peptide)

INTERVENTIONS:
Drug: CD-NP (Chimeric natriuretic peptide) — Infusion of CDNP at two of four doses

SUMMARY:
To access the efficacy of intravenous (IV) administration of CD-NP on changes in cardiac output and wedge pressure in patients with stabilized acute heart failure

ELIGIBILITY:
Key Inclusion Criteria:

* Hospitalization for AHF
* In need of hemodynamic monitoring

Key Exclusion Criteria:

* Administration of intravenous radiographic contrast agent within 7 days prior to screening or planned IV contrast media administration in the 4 days after screening or acute contrast-induced nephropathy at the time of screening
* Current or planned treatment with any IV therapies, including diuretics, vasodilators (including nesiritide), vasopressin antagonists, positive inotropic agents and vasopressors, or mechanical support
* Current or planned ultrafiltration, hemofiltration, or dialysis within 7 days of screening
* Significant pulmonary disease
* Known valvular heart disease
* Any organ transplant recipient or patient currently listed for transplant or admitted for any transplantation.
* Major surgery within 30 days of screening
* Other major disability or disease with expected survival less than 6 months.
* Major neurologic event, including cerebrovascular events, in the 60 days prior to screening
* Clinical diagnosis of acute coronary syndrome within 45 days of screening
* Troponin T ≥ 3 times the upper limit of normal at screening
* Significant arrhythmias
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy
* Liver function abnormality
* Administration of an investigational drug or implantation of investigational device, or participation in another trial, within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac output and wedge pressure | 8 hours

SECONDARY OUTCOMES:
Changes in additional hemodynamic measures | 8 hours
Diuresis and natriuresis during and after administration of study drug | 36 hour
Safety of CD-NP | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao Lieu, MD, Study Director — Nile Therapeutics Inc.; Gad Cotter, MD, Study Director — Momentum Research, Inc.
Locations (1):
- Russian Academy of Medical Sciences, Moscow, Russia, Russia